CLINICAL TRIAL: NCT04519632
Title: End-of-Life Pain Management by Carers and Healthcare Professionals in Infants, Children and Young People in Out of Hospital Settings
Brief Title: Paediatric Palliative Care Pain Management in the Community
Acronym: PARAMOUNT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Southampton (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Alder Hey Children's NHS Foundation Trust (Other); Helen & Douglas House Hospice, Oxford, UK (Unknown); Rainbow Hospice (Other)
Responsible Party: Sponsor
Other Study IDs: 47244
Record Dates: First submitted 2019-06-27; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Palliative Medicine; Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parents: Qualitative interviews
  Interventions: Other: Qualitative study
- Healthcare Professionals: Qualitative interviews
  Interventions: Other: Qualitative study
- Children: Children and young people aged 6-18 years, Qualitative interviews
  Interventions: Other: Qualitative study

INTERVENTIONS:
Other: Qualitative study — Qualitative interviews

SUMMARY:
To describe the the barriers and facilitators experienced by carers and healthcare professionals when managing medicines for pain relief for infants, children, and young people approaching the end of life in out of hospital settings.

DETAILED DESCRIPTION:
This study aims to hear about the experiences of patients, carers and healthcare professionals when managing pain relief medicines for infants, children and young people (ICYP) at the end of their lives, when they are not in hospital.

The study plans to develop a guide to help educate and empower both carers and healthcare professionals in the best ways to manage pain in this group of patients. This guide will contain basic, easily understood information depending upon both the patient's and carers' needs. Family carers are important in looking after their ICYP with life-threatening illnesses, so they can be cared for at home if they wish. Even with varying levels of support from hospice, hospital or family doctors, such responsibility can be rewarding and scary.

Community based healthcare professionals often have little experience to be able to support good end of life pain care in these patients when at home and there may be problems which prevent them from giving effective treatment. If pain and other symptoms are not well controlled by medicines families often move from their chosen place of care. Carers need to be able to check symptoms to decide which medicines to give and how well they are working, without having any special training; some may have unhelpful views about medicines such as morphine.

Not much research has looked at the problems that carers and healthcare professionals come across when trying to manage a child's pain when they are not in hospital.

Research has already shown that being able to provide the right medicine at the right time means children can be looked after where they want, without unnecessary hospital admissions. It is hoped that the guide will make carers feel more confident in managing pain relief safely, so lessening any worries. Future research is planned to show the value of the guide in a larger study.

ELIGIBILITY:
Inclusion Criteria

* Carers of infants, children, and young people up to 18 years being cared for outside hospital at the end of life (defined as those patients who score as 'orange' or 'red' on the Spectrum of Palliative Care Needs tool and/or who have a symptom management plan (including pain management) written by a specialist palliative care team.
* Self-reported full or partial responsibility for managing the patient's medicines, in particular having to select PRN (pro re nata or 'taken as needed') for pain and being responsible for the clinical decision making and the physical process of administering medicines.
* Healthcare professionals in primary, secondary and tertiary care who are involved in the care of children at end-of-life (defined as those patients who score as 'orange' or 'red' on the Spectrum of Palliative Care Needs tool) outside hospital, some of whom may be caring for the families taking part.
* Children and young people aged 6-18 years who are being cared for outside hospital at the end of life defined as those patients who score as 'orange' or 'red' on the Spectrum of Palliative Care Needs tool).

Exclusion Criteria:

* Carers judged by consultants or nurses to lack capacity to consent.
* Carers judged by nurses to be 'struggling' too much (however, these carers will still be able to approach the researcher directly if they wish to take part as posters will be used to advertise the study).
* CYP judged by carers or nurses to lack capacity to take part in an interview, who are too unwell or those who might find it too distressing.

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents and carers of infants, children and young people at the end-of-life being cared for in the community, the healthcare professionals supporting them, and the children and young people who receive this care
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative data obtained from semi-structured interviews | Baseline
  Barriers and facilitators to managing pain in infants, children, and young people at end of life as reported by parents, caregivers, healthcare professionals and children and young people.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Liossi, PhD, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided